CLINICAL TRIAL: NCT06290700
Title: Effect of Neonatal Care Education for Primiparous Pregnant Women on Postpartum Maternal Function and Quality of Life: Randomised Controlled Trial
Brief Title: Effect of Neonatal Care Education for Primiparous Pregnant Women on Postpartum Maternal Function and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCBU_2880
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Life Quality; Functional Status
Keywords: functional status; life quality; mothers; Pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervational group (Experimental): Neonatal care education given to primiparous pregnant women affect their postpartum maternal function Neonatal care education given to primiparous pregnant women affect their postpartum quality of life?
  Interventions: Behavioral: Neonatal Care education
- Control group (No Intervention): All pregnant women, those in the control group, were provide with standard

INTERVENTIONS:
Behavioral: Neonatal Care education — Participants who met the study inclusion criteria were provided with information about the purpose and conduct of the study, and their consent to participate was then obtained. The interviews were conducted in the breastfeeding room at the Uşak Dikilitaş Family Health Centre. The data were collected between November 2022 and November 2023. The Family Health Centre has two vaccination rooms, two antenatal care rooms, two observation rooms, and two breastfeeding rooms. Each pregnant woman was individually enrolled in an education session held in the breastfeeding room. The breastfeeding room was approximately 20 m², which was considered standard for accommodating training for an average of three pregnant women. The breastfeeding room was quiet, had a suitable temperature, and was located on the first floor in the middle of the corridor.
  Arms: İntervational group

SUMMARY:
This study aimed to evaluate the effect of neonatal care education for primiparous pregnant women on postpartum maternal function and quality of life.

DETAILED DESCRIPTION:
This was a single blind randomised controlled experimental study. The sample size of the study was calculated using the G*Power 3.1.7 program, considering a 5% margin of error and 95% confidence interval, and was determined to be at least 61. Therefore, the sample was planned to consist of 122 pregnant women, including 61 pregnant women in the intervention group and 61 pregnant women in the control group.

Study Inclusion Criteria Being at least a primary school graduate. Being a primiparous pregnant woman. Being able to provide feedback. Study Exclusion Criteria Being a multiparous pregnant woman. Being a high-risk pregnant woman. Participants who met the study inclusion criteria were provided with information about the purpose and conduct of the study, and their consent to participate was then obtained. The interviews were conducted in the breastfeeding room at the Uşak Dikilitaş Family Health Centre. The data were collected between November 2022 and November 2023. The Family Health Centre has two vaccination rooms, two antenatal care rooms, two observation rooms, and two breastfeeding rooms. Each pregnant woman was individually enrolled in an education session held in the breastfeeding room. The breastfeeding room was approximately 20 m², which was considered standard for accommodating training for an average of three pregnant women. The breastfeeding room was quiet, had a suitable temperature, and was located on the first floor in the middle of the corridor.

ELIGIBILITY:
Inclusion Criteria:

* Being at least a primary school graduate.
* Being a primiparous pregnant woman.
* Being able to provide feedback.

Exclusion Criteria:

* Being a multiparous pregnant woman.
* Being a high-risk pregnant woman.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
severity of maternal function by Barkin Index of Maternal Functioning | 10 weeks after after the intervention
  The scale was used 6 weeks after childbirth

SECONDARY OUTCOMES:
Maternal Postpartum Quality of Life Instrument | 10 weeks after after the intervention
  The scale was used 6 weeks after childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Yonca ÇIÇEK OKUYAN, Manisa, Turkey (Türkiye)